CLINICAL TRIAL: NCT02788292
Title: Effect of N-Acetylcysteine on Autologous Fat Graft Survival
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to hire research staff
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1021326
Record Dates: First submitted 2016-04-18; First posted 2016-06-02 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-10

CONDITIONS: Adipose Tissue Atrophy; Deformity of Reconstructed Breast; Graft Loss
Keywords: acetylcysteine; three-dimensional reconstruction; autologous fat grafting
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetylcysteine (NAC) (Experimental): NAC added to tumescent solution for liposuction and eventual fat grafting.
  Interventions: Drug: Acetylcysteine
- Control (No Intervention): Just tumescent solution for liposuction and fat grafting.

INTERVENTIONS:
Drug: Acetylcysteine — See arm description
  Other Names: N-acetylcysteine
  Arms: Acetylcysteine (NAC)

SUMMARY:
A single-centre triple-blind study looking at the addition of NAC to tumescent solution for liposuction and fat grafting in healthy patient volunteers already undergoing bilateral breast reduction. Three-dimensional reconstructions and volumetric analysis will be performed based on CT scans at 0, 1 and 3 months and then histological analysis will be performed after fat graft explantation at 3 months to determine fat graft vascularity and quality.

DETAILED DESCRIPTION:
Autologous fat grafting is an increasingly popular technique for soft tissue reconstruction; however, the surgical technique is limited by inconsistent graft take, undercorrection, and requirement for repeat procedures. The authors previously examined whether a widely available, clinically safe anti-oxidant, N-acetylcysteine (NAC), could improve adipose-derived stem cell survival and subsequent graft take when added to tumescent solution at the time of fat harvest in mice. The addition of NAC to tumescent fluid during fat harvest in mice protects ADSCs against oxidative stress, increases their survival and proliferation, and inhibits their early differentiation into mature adipocytes in vitro. In an in vivo model, NAC treatment at the time of harvest improved survival and quality of autologous fat grafts. These observations provide proof-of-principle for the use of NAC in the clinical setting to optimize fat graft yields.

Hypothesis: The addition of NAC to the tumescent solution used in fat grafting will improve fat graft survival in humans to potentially decrease the amount of re-operations and undercorrection that occurs.

Plan: The study will be conducted as a single-centre, randomized, triple-blind placebo-controlled trial to be performed at the QEII Health Sciences Centre, Halifax, Nova Scotia. Subjects will be chosen as healthy female patients already presenting to the operating room for elective breast reduction surgery. These patients will be enrolled and booked for surgery as they present to clinic and will not be expedited in receiving their elective surgery if enrolled in the study. Each subject will serve as her own control. The hypothesis will be tested by performing lipoaspiration of the thigh/hip region of healthy patients after the addition of tumescent solution with or without NAC. Approximately 10 millilitres of the fat graft will be injected into each pre-tibial area depending on the randomization allocation, as described by Kolle et al. (1) The volume of fat graft will be measured at 0, 1 and 3 months using computed tomographic (CT) scans according to institutional standards. The CT images will be exported into Materialise Interactive Medical Image Control System (MIMICS) and volumetric three-dimensional reconstructions will be made to measure the size and volume of the grafts at each of the time points. The grafts will then be explanted at 3 months and weighed. The histologic appearance, graded on the amount of inflammation, cysts/vacuoles, integrity and vascularity with CD31 staining will be assessed. The results will be compared using two-tailed t-tests. Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Women
2. Desire and surgical indication for liposuction of the thigh/hip region for women already undergoing elective breast reduction surgery
3. Age 18-45 years
4. BMI of 20-30
5. ASA Class I

Exclusion Criteria:

1. Known chronic illnesses: Diabetes, HIV, renal/liver failure, metabolic disease, history of cancer or family pre-disposition of cancer, peripheral vascular disease, illness that would preclude a general anaesthetic
2. Pregnancy or planned pregnancy within 1 year
3. Contraindications to CT
4. Previous hip/thigh surgery or injury
5. Previous lower leg surgery/injury
6. Smoker
7. Breastfeeding
8. Other disease according to investigator's judgment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Change in fat graft volume over time | 0, 1 and 3 months
  Based on CT scans of fat grafts and three-dimensional reconstructions/volumetric analysis

SECONDARY OUTCOMES:
Weight of fat graft | 3 months
  Fat grafts will be explanted and weighed at 3 months.
Fat graft vascularity | 3 months
  Vascularity of fat graft with CD31 staining.
Fat graft quality | 3 months
  Quality of fat graft through histological analysis of cysts/vacuoles/intact fat cells/fibrosis and also through adipocyte slide coverage analysis.
Adverse effects or complications | 1 year
  Collecting data regarding any adverse complications of the fat grafting procedure and subsequent recovery.

IPD SHARING:
Plan to Share IPD: No
IPD will not be available, but will be published as an average of outcomes.